CLINICAL TRIAL: NCT06811116
Title: A Phase I/II Trial of Sapanisertib in Combination With Cabozantinib in β-catenin-mutated Hepatocellular Carcinoma (SAPHIRE)
Brief Title: Testing the Addition of an Anti-cancer Drug, Sapanisertib, to the Usual Chemotherapy Treatment (Cabozantinib) in Metastatic Liver Cell Cancer With a Change in Genes for the Protein β-Catenin, The SAPHIRE Trial
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2025-00837; NCI-2025-00837 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 25-082; 10703 (Other: UPMC Hillman Cancer Center LAO); 10703 (Other: CTEP); UM1CA186690 (NIH)
Record Dates: First submitted 2025-02-05; First posted 2025-02-06 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Advanced Hepatocellular Carcinoma; Metastatic Hepatocellular Carcinoma; Stage III Hepatocellular Carcinoma AJCC v8; Stage IV Hepatocellular Carcinoma AJCC v8
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Specimen Handling; cabozantinib; X-Rays; sapanisertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (Sapanisertib + cabozantinib) (Experimental): Patients receive sapanisertib PO QD on 3 days on and 4 days off per week, 5 days on and 2 days off per week or on days 1-28 of each cycle and cabozantinib PO QD on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo blood collection and imaging scans throughout the study.
  Interventions: Procedure: Biospecimen Collection; Drug: Cabozantinib S-malate; Procedure: Imaging Procedure; Drug: Sapanisertib
- Arm II (Cabozantinib) (Active Comparator): Patients receive cabozantinib PO QD on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo blood collection imaging scans throughout the study.
  Interventions: Procedure: Biospecimen Collection; Drug: Cabozantinib S-malate; Procedure: Imaging Procedure

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Cabozantinib S-malate — Given PO
  Other Names: BMS-907351; Cabometyx; Cometriq; XL 184; XL-184; XL184
Procedure: Imaging Procedure — Undergo imaging scans
  Other Names: Diagnostic Imaging Technique; Image Type; Imaging; Imaging (procedure); Imaging Procedures; Imaging Technique; imaging type; IMAGING_METHOD; imaging_type; Medical Imaging; Type of imaging
Drug: Sapanisertib — Given orally (PO)
  Other Names: INK-128; INK128; MLN-0128; MLN0128; TAK-228
  Arms: Arm I (Sapanisertib + cabozantinib)

SUMMARY:
This phase I/II trial studies the side effects and best dose of sapanisertib when given together with cabozantinib, and to see how well they work in treating patients with liver cancer that has spread from where it first started to other places in the body (metastatic) and contains a mutation (change) in the β-catenin gene. Sapanisertib and cabozantinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving sapanisertib and cabozantinib together may work better than giving cabozantinib alone in treating β-catenin-mutated metastatic hepatocellular carcinoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To establish the recommended phase 2 dose (RP2D) of the combination of sapanisertib and cabozantinib in advanced hepatocellular carcinoma (HCC) patients. (Safety Lead-In [Phase I]) II. To determine the activity by progression free survival (PFS) of the combination of sapanisertib and cabozantinib versus (vs) cabozantinib alone in advanced β-catenin mutated HCC patients. (Phase II)

SECONDARY OBJECTIVES:

I. To estimate the activity by objective response rate (ORR) of the combination of sapanisertib and cabozantinib versus cabozantinib alone in advanced β-catenin mutated HCC patients.

II. To determine the activity by overall survival (OS) of the combination of sapanisertib and cabozantinib vs cabozantinib alone in advanced β-catenin mutated HCC patients.

III. To determine the safety and tolerability of the combination of sapanisertib and cabozantinib.

IV. To identify molecular subpopulations associated with response. V. To explore the pharmacokinetics (PK) for sapanisertib and cabozantinib.

EXPLORATORY OBJECTIVES:

I. To identify ribonucleic acid (RNA) signatures associated with response. II. To evaluate circulating tumor DNA (ctDNA) as a predictor for treatment response to therapy.

III. To explore the exposure response relationships for sapanisertib and cabozantinib.

OUTLINE: This is a phase I, dose-escalation study of sapanisertib and cabozantinib followed by a phase II randomized study. Patients in Phase I receive treatment as in Arm I. Patients in Phase II are randomized to 1 of 2 arms.

ARM I: Patients receive sapanisertib orally (PO) once daily (QD) on 3 days on and 4 days off per week, 5 days on and 2 days off per week or on days 1-28 of each cycle and cabozantinib PO QD on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo blood collection and imaging scans throughout the study.

ARM II: Patients receive cabozantinib PO QD on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo blood collection imaging scans throughout the study.

After completion of study treatment, patients are followed up every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed HCC, not amenable to curative treatment approach
* For Phase 2, patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as ≥ 20 mm (≥ 2 cm) by chest x-ray or as ≥ 10 mm (≥ 1 cm) with CT scan, MRI, or calipers by clinical exam
* For phase 2, patients must have a β-catenin mutation, based on next generation eequencing (NGS) testing through Clinical Laboratory Improvement Amendments (CLIA)-certified commercially available standard of care assay
* Patients must have received at least one prior line of systemic therapy in the metastatic setting, including a prior immune checkpoint inhibitor therapy unless not eligible. For the phase 2 portion, patients must have received at least one and no more than two prior lines of systemic therapy in the metastatic setting, including a prior immune checkpoint inhibitor therapy unless not eligible
* Age ≥ 18 years. Because no dosing or adverse event data are currently available on the use of sapanisertib in combination with cabozantinib in patients <18 years of age, children are excluded from this study
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 (Karnofsky ≥ 50%)
* Child Pugh score of A
* Absolute neutrophil count ≥ 1,000/mcL
* Platelets ≥ 30,000/mcL
* Total bilirubin ≤ 1.5 × institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT)(serum glutamic pyruvic transaminase [SGPT]) ≤ 5 × institutional ULN
* Glomerular filtration rate (eGFR) ≥ 40 mL/min/1.73 m^2
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression
* Patients with new or progressive brain metastases (active brain metastases) or leptomeningeal disease are eligible if the treating physician determines that immediate CNS specific treatment is not required and is unlikely to be required during the first cycle of therapy
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class II or better
* For the phase 2 portion, availability of archival tumor tissue at the time of patient enrollment for banking for molecular profiling studies
* The effects of sapanisertib and cabozantinib on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and after completion of drug administration. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Both men and women treated or enrolled on this protocol must agree to use adequate contraception prior to the study, for the duration of study participation, and for the following duration after completion of sapanisertib and cabozantinib administration:

  * 90 days and 120 days after last dose of sapanisertib for women of childbearing potential and men respectively,
  * 5 months and 7 months after last dose of cabozantinib for women of childbearing potential and men respectively
* Ability to understand and the willingness to sign a written informed consent document. Legally authorized representatives may sign and give informed consent on behalf of study participants

Exclusion Criteria:

* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1) with the exception of alopecia
* Patients who are receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to sapanisertib and cabozantinib
* Use of strong CYP3A4-inhibiting agents due to drug-drug interaction with cabozantinib
* Prior exposure to cabozantinib
* Patients who are unable to swallow oral medications such as capsules and tablets and patients with gastrointestinal conditions that may affect the absorption of oral medications
* Patients with uncontrolled intercurrent illness or any other significant condition(s) that would make participation in this protocol unreasonably hazardous
* Pregnant women are excluded from this study because sapanisertib and cabozantinib have the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with sapanisertib and cabozantinib, breastfeeding should be discontinued if the mother is treated with sapanisertib and cabozantinib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2025-11-17 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicities and incidence of adverse events | From registration to disease progression or death due to any cause, assessed up to 2 years
  Dose limiting toxicities and adverse events per Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 will be tabulated for each dose level.
Progression free survival (PFS) | From registration to disease progression or death due to any cause, assessed up to 2 years
  Treatment response will be assessed based on Response Evaluation Criteria in Solid Tumors version 1.1. PFS will be estimated by the Kaplan-Meier method, along with 95% confidence regions. Median PFS will also be calculated along with its 95% confidence intervals (CI).

SECONDARY OUTCOMES:
Objective response rate (ORR) | From registration to disease progression or death due to any cause, assessed up to 2 years
  Defined as the proportion of patients with complete response or partial response. ORR will be estimated along with its exact 95% CI.
Overall survival (OS) | From registration to disease progression or death due to any cause, assessed up to 2 years
  Will be estimated by the Kaplan-Meier method, along with 95% confidence regions. Median OS will also be calculated along with its 95% CI.
Incidence of adverse events | Baseline up to 2 years
  Will be tabulated according to CTCAE version 5.0 type, grade and relation to treatment in combination and in the control arm. The worst grade of adverse event will be determined for each participant
Whole exome sequencing on archival tissue | At pre-treatment for phase II
  Mutations with a focus on the MET pathway; TERT promoter mutations, NEFL2; TSC1/2; TERT; ARID1a; ARID2; CTNNB1; TP53; AXIN1-2, APOB, ALB, MLL2, and others as well as somatic mutation burden will be assessed in archival tissue and we will evaluate any relations with peculiar response.
Sapanisertib and cabozantinib pharmacokinetics (PK) | From pre dose on cycle 1 day 8 to pre dose on cycle 3 day 1 for phase I and II
  Sapanisertib and cabozantinib exposure will be described and compared to historical controls

OTHER OUTCOMES:
Tumor signatures in archival bulk RNAseq | During phase II
  For mTOR, Met and NRF2. After correction for batch effect (limma R package), gene set variation analysis scores for each gene set described will be calculated for each patient tumor sample. For sapanisertib, we propose to use 19-gene signature as well as 28-gene signature previously identified as a biomarker of Nrf2 pathway activation and used by us. For cabozantinib, we will be using signatures derived from KAPOSI_LIVER_CANCER_MET_UP" consisting of 18 genes which we have used earlier. We will evaluate any relations with peculiar response.
Change in variant allele frequencies (VAF) of tumor mutations in circulating tumor-derived deoxyribonucleic acid (DNA) (ctDNA) | Pre-treatment to cycle 3
  The detectable VAFs will be assessed and trended during the course of treatment. VAF change will be assessed categorically for each patient (increased or decreased at cycle 3 as compared to pre-treatment). The association of VAF change with objective response will be tested using the Fisher's test, where p<0.05 will be considered statistically significant
Sapanisertib and cabozantinib PK and toxicity/response | From pre dose on cycle 1 day 8 to pre dose on cycle 3 day 1 for phase I and II
  Sapanisertib and cabozantinib exposure will be exploratorily correlated with toxicity and response with non-parametric tests at a significance level of 0.05 (PK endpoints in patients with vs without presence of toxicity or response endpoints). Cabozantinib PK as single agent versus in combination with sapanisertib will be compared with a paired non-parametric test at a significance level of 0.05

CONTACTS AND LOCATIONS:
Overall Officials: Anwaar Saeed, Principal Investigator — UPMC Hillman Cancer Center LAO
Locations (4):
- United States (4):
  - UCI Health - Chao Family Comprehensive Cancer Center and Ambulatory Care, Irvine, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Oregon Health and Science University, Portland, Oregon
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm